CLINICAL TRIAL: NCT06426030
Title: Validation of Czech Language Versions of Questionnaires Most Frequently Used for Functional Status Monitoring in Patients With Amyotrophic Lateral Sclerosis and the Long-term Follow-up of Biomarkers of the Disease in These Patients.
Brief Title: Validation of Czech Language Versions of Questionnaires for ALS Patients' Functional Status and Biomarker Long-term Follow-up
Status: Recruiting | Type: Observational
Sponsor: Masaryk University (Other)
Collaborators: Brno University Hospital (Other); University Hospital, Motol (Other); University Hospital, Martin (Other); University Hospital Bratislava (Other)
Responsible Party: Sponsor
Other Study IDs: VALID-ALS-QUEST-CZ
Record Dates: First submitted 2024-05-17; First posted 2024-05-23 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-05

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: Amyotrophic lateral sclerosis; ALS; ALSFRS-R; ALSFRS-EX; ALSAQ-40; Borg scale; Frontal assessment battery; Scale; Questionnaire
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Questionnaires and scales used to assess the clinical status and quality of life of patients with amyotrophic lateral sclerosis (ALS) are an important tool to monitor the disease progression and current needs of patients. The use of these tools (and in particular their combination) allows to cover the whole spectrum of potential patient difficulties and thus significantly facilitates the process of individualisation and optimisation of care. The aim of the study was to create and validate the Czech language versions of the following questionnaires or scales: (1) ALSFRS-R (ALS Functional Rating Scale - Revised Version) and (2) ALSFRS-EX (EXtended, i.e. extended, version of the same scale), both in the self-assessment version (incl. (3) the ALSAQ-40 (ALS Assessment Questionnaire including 40 questions), (4) the DYALS (Dysphagia in ALS), and (5) the Borg Dyspnoea Rating Scale.

All questionnaires were translated using the forward-backward translation method. The scales and questionnaires were administered to ALS patients repeatedly at one-week intervals, first in writing during routine patient follow-up at the Neuromuscular Centre of the University Hospital Brno, and during repeated administrations by telephone.

DETAILED DESCRIPTION:
The first step of the study (before patient recruitment began) was the linguistic validation of all the scales and questionnaires used. Initially, Czech language versions were created using the forward-backward translation method. These created versions were then discussed by an expert panel consisting of 2 amyotrophic lateral sclerosis experts and 2 translators (one native speaker bilingual for both Czech and English, one professional translator specialized in medical English).

Patients potentially meeting the entry criteria will be informed about the purpose and conduct of the study and will sign an informed consent if they agree to participate in the study.

The first administration of all questionnaires (including the self-assessment version of the ALSFRS-R, ALSFRS-Ex, ALSAQ-40, DYALS and Borg Scale for lying, standing and moving positions) will be performed as part of the patient's routine clinical follow-up at the neuromuscular centre. The other two administrations of the questionnaires will be done by telephone one and two weeks after inclusion, respectively. The one-week interval was chosen in line with the approach of similar foreign validation studies of other languages, so that there is a high probability of no significant change in the patient's clinical condition between repeated administrations and, on the other hand, that the patient no longer remembers in detail the answers from the previous administration. At the first telephone readministration (after one week), patients will complete the full range of questionnaires as they did at the first administration of the questionnaires at the centre. The second telephone readministration (after an additional week) will involve completion of the ALSFRS-R and -EX questionnaires only and will use the standard version of both questionnaires administered by an assessor certified to use this scale.

For patients with significantly limited verbal communication skills, it is acceptable to have the patient's caregiver mediate the responses during the telephone administration and/or to send the completed questionnaires during the follow-up administrations by mail or electronically (e-mail). In these cases, patients will be invited to complete the readministration questionnaires by email or telephone (depending on their preference) at a time that would be consistent with normal telephone readministrations for other patients (to maintain an identical time interval between readministrations). Similarly, for patients with limited ability to grasp writing instruments, it will be permissible to complete questionnaires in collaboration with the caregiver, but always on the basis of patient-reported data.

At the first administration of all questionnaires (including the self-assessment version of the ALSFRS-R questionnaire) at the centre, the patient will be asked to complete the questionnaires without further clarification from the investigator. Similarly, during the first telephone readministration involving only the self-assessment questionnaires, the individual questions and the options included in them will be read to the patient only, with no opportunity for the patient to ask additional questions, in order to maintain the self-assessment nature of all tests used.

The standard (non-self-assessment) version of the ALSFRS-R questionnaire will be administered at the second telephone follow-up by TRICALS (Treatment Research Initiative to Cure ALS, an organisation authorised to use the questionnaire in a certified manner) certified assessors and will be administered in accordance with the training provided by this initiative. Initial and repeat administrations will be conducted by different raters. Evaluators conducting telephone readministrations will not be aware of patients' initial test results at the first administration or their clinical status.

The procedures for working with human subjects were approved by the Ethics Committee of the Brno University Hospital on 11.05.2023, reference number 06-110522/EK, project number 85/22.

Statistical data processing will be performed using SPSS 29 statistical software (IBM Corporation, 2020, Armonk, New York, USA).

ELIGIBILITY:
Inclusion Criteria:

1. diagnosed amyotrophic lateral sclerosis (ALS) meeting the EMG (electromyographic) criteria:

   * Gold Coast criteria or
   * at least clinically probable ALS according to Awaji-Shima criteria
2. willing and able to comply with all protocol procedures

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: ALS patients in colaborating Centres - University Hospital Brno (CZ), Motol University Hospital (CZ), Martin University Hospital (SK), University Hospital Bratislava (SK) - who are willing to participate in study.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-05-17 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Questionnaire validity (ALSFRS-R(-EX), ALSAQ-40, DYALS) | 01.09.2024
  Content Validity: Ensures the questionnaire comprehensively covers the construct it intends to measure.
Questionnaire reproducibility (Czech versions of ALSFRS-R(-EX), ALSAQ-40, DYALS) | 01.09.2024
  Test-Retest Reliability:
  Intraclass Correlation Coefficient (ICC) Pearson or Spearman Correlation Coefficient Cohen's Kappa (κ) Bland-Altman Plot
Agreement between self reported and non-self reported version of ALSFRS-R | 01.09.2024
  Test-Retest Reliability:
  Intraclass Correlation Coefficient (ICC) Pearson or Spearman Correlation Coefficient Cohen's Kappa (κ) Bland-Altman Plot

CONTACTS AND LOCATIONS:
Overall Officials: Eva Vlckova, doc,MD,PhD, Study Chair — Masaryk University, University Hospital Brno.
Locations (1):
- University Hospital Brno, Brno, Czech Republic, Czechia

IPD SHARING:
Plan to Share IPD: Undecided